CLINICAL TRIAL: NCT03879213
Title: The Effects of Acute Raspberry Intake on the Relationship Between Enhanced Metabolic Control and Cognitive and Psychomotor Function
Brief Title: Acute Berry Intake on Metabolic Control and Cognitive Function
Acronym: RRB3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB2018-046
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Raspberry; Metabolic responses; Endothelial function; Cognitive function

STUDY DESIGN:
Intervention Model Description: Multi center, randomized, single-blind, 2-arm, placebo-controlled, within subject cross-over trial, featuring a repeated postprandial sampling paradigm
Who Masked: Participant
Masking Description: Single (Participant) Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): freeze-dried red raspberry powder (25 g) in active breakfast meal
  Interventions: Dietary Supplement: Active breakfast
- Placebo (Placebo Comparator): Placebo breakfast
  Interventions: Dietary Supplement: Control breakfast

INTERVENTIONS:
Dietary Supplement: Active breakfast — freeze-dried red raspberry powder (12.5 g) in drink+ freeze-dried red raspberry powder (12.5 g) in buttermilk biscuit sandwich
  Arms: Active
Dietary Supplement: Control breakfast — Control drink + buttermilk biscuit sandwich
  Arms: Placebo

SUMMARY:
The objectives of this study are:

1. Evaluate the effects of acute dietary raspberry intake on metabolic-associated impairments in cognitive and psychomotor function in overweight/obese adults (55-70y) following a meal challenge
2. Evaluate the effects of acute dietary raspberry on measures of vascular function.

DETAILED DESCRIPTION:
The proposed study will be conducted in humans according to Good Clinical Practice (GCP) guidelines. All subjects will review and sign an Informed Consent Form approved by the Illinois Institute of Technology's Institutional Review Boards (IRB) prior to screening.

This multi-center clinical trial is a randomized, single-blind, 2-arm, placebo-controlled, within subject cross-over trial, featuring a repeated postprandial sampling paradigm to evaluate the effects of acute dietary red raspberry intake on cognitive function, inflammation, insulin sensitivity / glucose handling and vascular function in overweight/obese older adults after consuming a standardized challenge meal.

A planned sample size of 30 will be enrolled into the study. This study will require one initial screening visit and 3 study visits. This study will take approximately 3-4 weeks per subject to complete.

The initial screening visit will provide subject with their site-specific, IRB-approved informed consent document prior to the start of any study related procedures. Subject eligibility will be determined through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey relate to general eating, health, mood and exercise habits.

Eligible subjects will follow a limited polyphenolic diet throughout the duration of their participation, although stricter guidelines will be imposed during the 3 days prior to a study visit. Shopping lists and meal plans will be provided to subjects, along with counseling by the investigator's study dietitians, to help subjects adhere to the limited polyphenolic diet. The trial will initiate with a 3-day food diary to assess background (pre-study) dietary intake followed by counseling to follow a diet relatively low in (poly)phenolic rich-beverages/foods, which will be maintained for the duration of the experiment. After an initial 7 day run-in period on the limited polyphenolic diet, subjects will be randomized to 1 of 2 treatment sequences. Treatment codes will be maintained by the principal investigator/study physician. All subjects will receive both treatments, once each on 2 different occasions and separated by at least 1 week. Red raspberries or placebo will be provided with a standardized meal providing 840 kcal. A low-polyphenol snack will be provided to subjects after their final cognitive assessment.

Each visit will last ~ 9.5 hours and subjects will be required to remain at the Clinical Unit for the duration of the visit. Blood samples will be collected at 0 (fasting) and at 0.5 h, 1 h, 2 h, 4 h, 5 h, 6 h and 7.5 h via a catheter placed on the non-dominant arm by a registered nurse. Cognitive function will be measured at 0 (fasting), 2 h, and 6 h. FMD or NIRS will be conducted at the CNRC or the HNRCA, respectively at 0 (fasting), and at 1 h and 5 h.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27 and 35 kg/m2 and/or waist circumference (>35 inches for women, >40 inches for men)
* Aged 55-70 years old
* Able to provide informed consent and comply with study procedures
* Willing to maintain stable body weight and follow his/her habitual diet and physical activity patterns throughout the trial.
* Judged by the Investigator to be in general good health on the basis of medical history and screening laboratory tests.

Exclusion Criteria:

* Current smoker and/or marijuana user, past smokers may be allowed in the study if stopped >2 years
* Have a history or presence of atherosclerotic cardiovascular disease, inflammatory disease, diabetes mellitus, or other systemic diseases, psychological or psychiatric disorders
* Have recent surgery or injury to head
* Mini-Mental Status Exam score < 24 or Beck Depression Inventory score > 20
* Taking any medications that would interfere with outcomes of the study (i.e., lipid-lowering medications, anti-inflammatory drugs, and supplements, not including multivitamin/mineral or calcium/Vit D supplements),
* Unstable use of any medication/supplement
* Have a history of cancer in the prior 5 years, except for non-melanoma skin cancer
* Addicted to drugs and/or alcohol (>2 drinks/day)
* Have been exposed to any non-registered drug product within last 30 days.
* Working overnight (e.g. 3rd shift of overnight workers)
* Excessive exercisers or trained athletes
* Have allergies/intolerances to berries.
* Vegetarian/vegan or have extreme dietary habits.
* Excessive coffee/tea drinker
* Actively losing weight/ trying to lose weight (unstable body weight fluctuations of > 5 kg in 3 months)
* Donated blood within last 3 months
* Female who is pregnant, planning to be pregnant, breastfeeding
* Current regular consumption of berries which exceeds > 2 servings per day
* The individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in Profile of Mood States response between 2 treatments | Baseline to 6 hours
  Cognitive assessment tasks will be performed in Profile of Mood States
Changes in Digit Symbol Coding response between 2 treatments | Baseline to 6 hours
  Cognitive assessment tasks will be performed in Digit Symbol Coding
Changes in Hopkins Verbal Learning Test response between 2 treatments | Baseline to 6 hours
  Cognitive assessment tasks will be performed in Hopkins Verbal Learning Test
Changes in CANTAB- paired-associates-learning response between 2 treatments | Baseline to 6 hours
  Cognitive assessment tasks will be performed in CANTAB- paired-associates-learning
Changes in CANTAB- rapid-visual-information-processing response between 2 treatments | Baseline to 6 hours
  Cognitive assessment tasks will be performed in CANTAB- rapid-visual-information-processing
Changes in CANTAB- spatial-working-memory response between 2 treatments | Baseline to 6 hours
  Cognitive assessment tasks will be performed in CANTAB- spatial-working-memory

SECONDARY OUTCOMES:
Changes in Psychomotor function between 2 treatments | Baseline to 6 hours
  Psychomotor function will be measured with the Grooved Pegboard
Changes in postprandial endothelial function between 2 treatments | Baseline to 5 hours
  Vascular Assessments will be measured with Flow mediated vasodilation (FMD)

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States